CLINICAL TRIAL: NCT07036887
Title: Effectiveness of 1st Rib Mobilization and Scalene Muscles Muscle Energy Technique Among Patients With Asthma
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall20/1001
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Rib Mobilization + Respiratory Physiotherapy (Experimental)
  Interventions: Diagnostic Test: First Rib Mobilization + Respiratory Physiotherapy
- Scalene Muscle Energy Technique (MET) + Respiratory Physiotherapy (Active Comparator)
  Interventions: Combination Product: Scalene Muscle Energy Technique (MET) + Respiratory Physiotherapy

INTERVENTIONS:
Diagnostic Test: First Rib Mobilization + Respiratory Physiotherapy — Patients were given post isometric relaxation for restricted first rib in sitting position and therefore the affected elevated first rib, opposite foot of therapist was placed on the table and patient non affected arm is 'dropped' on the therapist flexed knee. The practitioner's conjointly flexes the elbow on the non-affected side placed anterior to shoulder with the hand supporting the patient facet of head. Then therapist makes contact with the tubercle of the first rib with fingers or thumb of affected side (patient) disposing of available soft tissue. slack as steady force is applied in inferior direction. The therapist eases his flexed leg and uses his supported hand to encourage patient's neck into a side flexion and rotation to affected side thus unloading the scalene tension thereon side and encourage the first rib to move anteriorly and inferiorly
  Arms: First Rib Mobilization + Respiratory Physiotherapy
Combination Product: Scalene Muscle Energy Technique (MET) + Respiratory Physiotherapy — MET for the scalene muscle, the participants were made to lie supine with a cushion or towel under the upper thoracic area. The PT placed his hand on the side of the participant's face/forehead to resist the isometric contraction and the other hand on the sternum. The participants were asked to perform the action of the anterior scalene muscle against PT resistance and hold it for 7-8 seconds followed by relaxation. (42) Along with the same respiratory physiotherapy protocol used in Group A. The treatment protocol was given for three sessions per week for four weeks
  Arms: Scalene Muscle Energy Technique (MET) + Respiratory Physiotherapy

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of first rib mobilization and scalene muscle energy technique (MET) in improving respiratory function and reducing symptoms in patients with asthma. Asthma is a chronic inflammatory condition of the airways characterized by bronchoconstriction, airway hyperresponsiveness, and mucus overproduction, often leading to respiratory difficulty and increased use of accessory muscles such as the scalene.

DETAILED DESCRIPTION:
Manual therapy techniques like first rib mobilization and scalene MET are believed to restore upper thoracic mobility, reduce muscle tightness, and optimize breathing mechanics. In this study, 47 asthmatic patients will be randomly assigned into two groups: Group A will receive first rib mobilization combined with respiratory physiotherapy, while Group B will receive scalene MET along with the same physiotherapy protocol. Treatment will be administered three times a week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female age range: 18-65 years.
* Diagnosed with asthma according to the Global Initiative for Asthma criteria.
* Presence of musculoskeletal symptoms; Complaints of chest tightness, neck stiffness, or restricted upper thoracic mobility, often associated with dysfunctional breathing patterns.
* Ability to provide informed consent and comply with the treatment protocol.

Exclusion Criteria:

* clinically unstable or had a neuromuscular disease, unstable cardiovascular disease, or musculoskeletal disease that may interfere with exercise
* History of thoracic or cervical spine surgery, trauma, or fractures
* Pregnancy or postpartum status
* Rheumatologic diseases, a history of musculoskeletal trauma, or musculoskeletal malformations.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire (SGRQ) | 6 Month
  The total score has a maximum of 100 points, with values ranging from 0 to 100. The higher the number, the more impact the disease has.

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No